CLINICAL TRIAL: NCT02616887
Title: Phase II Study of Image-Guided Single Fraction SBRT With VMAT-FFF Technique for Vertebral Metastases
Brief Title: Study of Image-Guided SBRT for Vertebral Metastases
Status: Terminated | Type: Observational
Why Stopped: not sufficient patients enrolled
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, MD, Istituto Clinico Humanitas
Other Study IDs: 1460
Record Dates: First submitted 2015-11-24; First posted 2015-11-30 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Vertebral Metastases
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Vertebral metastases: Selected patients with spine metastases are treated with ablative single dose SBRT and VMAT technique in various solid tumors .
  Interventions: Radiation: Single dose SBRT and VMAT technique

INTERVENTIONS:
Radiation: Single dose SBRT and VMAT technique — One fraction of 18 Gy delivered in one day with VMAT and Flattening filter-free (FFF) beams.

SUMMARY:
Based on the known efficacy of ablative single dose SBRT and VMAT technique in various solid tumors, investigators have designed this study to assess feasibility of SBRT in selected patients with spine metastases.

DETAILED DESCRIPTION:
This is a prospective, phase 2 study. The main objectives are to assess acute and late side effects of single fraction SBRT for selected patients with vertebral metastases and to study the local control of disease in treated sites.

The schedule will be 1 fraction of 18 Gy delivered in one day with Volumetric Modulated Arc Therapy (VMAT) and Flattening filter-free (FFF) beams.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18years.
* WHO performance status ≤ 2 (ECOG - KPS).
* Histologically-proven of primary cancer disease.
* Metastatic disease in the spine, from C1 to Sacrum. A maximum number of 5 sites. Each of the separate sites may have a maximal involvement of 2 contiguous vertebral bodies.
* Epidural compression is eligible when there is at least 3 mm gap between the spinal cord and the edge of the epidural lesion, unless patient underwent decompression surgery.
* A paraspinal mass ≤ 5 cm.
* Minimal residual tumor after surgery
* Metastases in other district of the body are allowed.
* Informed consent.

Exclusion Criteria:

* > 50% loss of vertebral body height.
* Prior radiation to the interested spine.
* Patients for whom an MRI of the spine is medically contraindicated.
* Patients allergic to contrast used in MRIs or CT scans or who cannot be premedicated for the use of contrast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with spine metastases
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
Toxicity of single fraction SBRT on spine metastases using CTCAE v.4 | 1 year
Local control of the treated lesions using Kaplan-Meyer statistical curves | 1 year

SECONDARY OUTCOMES:
Pain control at treated sites after RT using CTCAE v.4 | 3 months
Local control of the metastatic disease using Kaplan-Meyer statistical curves | 3 months
Overall survival of treated patients using Kaplan-Meyer statistical curves | 1 year
Difference of local and pain control between patients operated on vertebra and non-operated patients using CTCAE v.4 | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Franzese, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy